CLINICAL TRIAL: NCT06208488
Title: A Phase 1, Open-label, Randomized, Parallel-group Study to Evaluate the Pharmacokinetics, Pharmacodynamics, Safety, Immunogenicity, and Device Performance of ALXN1720 (Gefurulimab) Administered Subcutaneously Using Prefilled Syringe Versus Autoinjector in Adult Healthy Participants
Brief Title: A Study of Subcutaneous Gefurulimab Using Prefilled Syringe Versus Autoinjector in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ALXN1720-HV-103
Record Dates: First submitted 2023-11-06; First posted 2024-01-17 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Healthy Adult Participants
Keywords: Pharmacokinetics; Pharmacodynamics; Safety; Immunogenicity; Device Performance

STUDY DESIGN:
Intervention Model Description: Separate randomization lists will be produced for each weight stratum (ie, 50 to < 70 kg, 70 to < 90 kg, and 90 to < 110 kg) and within each of the three weight strata, participants will be randomized 1:1:1:1:1:1 to one of the six combinations of device (PFS-SD or AI) and injection site (abdomen, thigh, or upper arm).
Who Masked: Outcomes Assessor
Masking Description: This is an open-label study. To avoid potential bias and maintain the data integrity, the analysis and reporting performed before database lock for Primary Analysis, ie, dry run/blinded data review for Primary Analysis, will be based on blinded data in which the treatment information is based on a dummy randomization schedule.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gefurulimab PFS-SD (Experimental): Participants will be administered gefurulimab as a single dose of 600 mg by PFS-SD on the abdomen, thigh, or upper arm.
  Interventions: Drug: Gefurulimab PFS-SD
- Gefurulimab AI (Experimental): Participants will be administered gefurulimab as a single dose of 600 mg by AI on the abdomen, thigh, or upper arm.
  Interventions: Drug: Gefurulimab AI

INTERVENTIONS:
Drug: Gefurulimab PFS-SD — Participants will receive a single 600 mg dose of Gefurulimab PFS-SD subcutaneously (SC) on Day 1.
  Other Names: ALXN1720
  Arms: Gefurulimab PFS-SD
Drug: Gefurulimab AI — Participants will receive a single 600 mg dose of Gefurulimab AI subcutaneously (SC) on Day 1.
  Other Names: ALXN1720
  Arms: Gefurulimab AI

SUMMARY:
This study will evaluate the pharmacokinetics (PK), pharmacodynamics (PD), safety, immunogenicity, and device performance of gefurulimab.

DETAILED DESCRIPTION:
This is an open-label, randomized, parallel-group study.

The study consists of 2 periods: a Screening Period (up to 70 days), and an Evaluation Period of 92 days.

Separate randomization lists will be produced for each weight stratum (50 to < 70 kg, 70 to < 90 kg, and 90 to < 110 kg) and within each of the three weight strata, participants will be randomized 1:1:1:1:1:1 to one of the six combinations of device (prefilled syringe with needle safety device [PFS-SD] or autoinjector [AI]) and injection site (abdomen, thigh, or upper arm),

Participants will receive a single dose of 600 mg gefurulimab on Day 1, will be residential at the clinical unit until Day 5, will have visits on Day 8, quaque week (once a week) [qw] thereafter until Day 50, and quaque 2 week (once every two weeks) [q2w] from Day 50 until Day 92 during the Evaluation Period.

The total study duration is up to 162 days.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be 18 to 65 years of age inclusive, at the time of signing the informed consent.
2. Body weight within ≥ 50 to < 110 kg and body mass index (BMI) within the range 18.5 to 30 kg/m2 (inclusive)
3. Participants who are healthy as determined by medical evaluation with no clinically significant or relevant abnormalities as determined by medical history, physical examination, vital signs, 12-lead ECG, and clinical laboratory evaluation.
4. QT interval corrected using Fridericia's formula (QTcF) ≤ 450 msec for male participants and ≤ 460 msec for female participants at Screening and prior to dosing on Day 1.
5. Documented vaccination against meningococcal infection from serogroups A, C, W, and Y and serogroup B.
6. Male and female participants should adhere to study-specific contraceptive methods.

Exclusion Criteria:

1. History of any Neisseria meningitidis infection.
2. History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrinological, hematological, or neurological disorders.
3. Abnormal blood pressure as determined by the Investigator.
4. History of latent or active TB (Tuberculosis) or exposure to endemic areas.
5. Allergy to monoclonal antibodies.
6. Clinically significant multiple or severe drug allergies, intolerance to topical corticosteroids, or severe posttreatment hypersensitivity reactions.
7. Lymphoma, leukemia, or any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years.
8. Current or chronic history of liver disease.
9. Known hepatic or biliary abnormalities.
10. Active systemic bacterial, viral, or fungal infection within 14 days prior to dosing.
11. History of allergy or intolerance to penicillin or cephalosporin.
12. History of clinically significant allergic reaction (eg, anaphylaxis or angioedema) to any product.
13. Live vaccine(s) within 1 month prior to Screening or plans to receive such vaccines during the study.
14. Evidence of human immunodeficiency virus (HIV) infection (positive HIV type 1 or type 2 antibody).
15. Evidence of hepatitis B infection (positive hepatitis B surface antigen [HBsAg] or positive total hepatitis B core antibody [HBcAb] with negative surface antibody [anti-HBs]), or hepatitis C viral infection (positive HCV RNA).
16. Female participants who have a positive pregnancy test at Screening or Admission.
17. Positive prestudy drug/alcohol screen; positive result may be repeated once.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2023-11-22 (Actual); Primary Completion 2024-09-17 (Actual); Study Completion 2024-09-28 (Actual)

PRIMARY OUTCOMES:
Area under the serum concentration-time curve from time zero to the last measurable concentration (AUClast) | Day 1 up to early discontinuation or Day 92
  The AUClast exposure in healthy participants following a single SC dose of 600 mg gefurulimab by AI comparable to the PK exposure using the PFS-SD will be assessed.
Area under the serum concentration-time curve from time zero to time infinity (AUCinf) | Day 1 up to early discontinuation or Day 92
  The AUClinf exposure in healthy participants following a single SC dose of 600 mg gefurulimab by AI comparable to the PK exposure using the PFS-SD will be assessed.
Maximum (peak) concentration observed after study intervention administration (Cmax) | Day 1 up to early discontinuation or Day 92
  The Cmax exposure in healthy participants following a single SC dose of 600 mg gefurulimab by AI comparable to the PK exposure using the PFS-SD will be assessed.

SECONDARY OUTCOMES:
Time to maximum observed serum concentration (tmax) | Day 1 to Day 92
  The tmax of gefurulimab SC in healthy participants across devices, and injection sites will be assessed.
Terminal elimination half-life (t½) | Day 1 to Day 92
  The t½ of gefurulimab SC in healthy participants across devices, and injection sites will be assessed.
Apparent total body clearance of the study intervention from serum (CL/F) | Day 1 to Day 92
  The CL/F of gefurulimab SC in healthy participants across devices, and injection sites will be assessed.
Apparent volume of distribution (Vd/F) | Day 1 to Day 92
  The Vd/F of gefurulimab SC in healthy participants across devices, and injection sites will be assessed.
Serum free C5 (complement component 5) concentrations | Day 1 to Day 92
  The serum free C5 concentrations of gefurulimab SC in healthy participants across devices and injection sites will be assessed.
Number of subjects with TEAEs (treatment-emergent adverse event) and TESAEs (treatment-emergent serious adverse event) | From Admission (Day-1) to Day 92
  The safety and tolerability of gefurulimab SC in healthy participants across devices and injection sites will be evaluated.
Incidence of antidrug antibody (ADA) to gefurulimab category of immune-response and titer | Day 1, Day 92
  The immunogenicity of gefurulimab SC administered with either PFS-SD or AI in healthy participants will be assessed.
Number of reported outcome of attempted full-dose administration via AI (autoinjector) or PFS-SD (prefilled syringe with needle safety device) | Day 1
  The performance of the AI and PFS-SD in the administration of gefurulimab SC in healthy participants will be assessed.
Number of reported device deficiencies/complaints and associated device investigations | Day 1
  The performance of the AI and PFS-SD in the administration of gefurulimab SC in healthy participants will be assessed.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Research Site, Toronto, Ontario
  - Research Site, Laval, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPINPhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/